CLINICAL TRIAL: NCT00653783
Title: Blood Alpha-Synuclein, Gene Expression, and Smell Testing as Diagnostic and Prognostic Biomarkers in Parkinson's Disease
Brief Title: Diagnostic and Prognostic Biomarkers in Parkinson Disease
Acronym: PROBE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: The Parkinson Study Group (Network)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Bernard Ravina, MD, MSCE, Principal Investigator, University of Rochester, Clinical Trials Coordination Center
Other Study IDs: U01NS050095-02_PROBE; DOD Grant # W81XWH-07-1-0007; NINDS Grant 5 U01 NS050095-02; U01NS050095-02 (NIH)
Record Dates: First submitted 2008-04-02; First posted 2008-04-07 (Estimated); Last update posted 2008-12-31 (Estimated); Status verified 2008-12

CONDITIONS: Parkinson Disease; Multiple System Atrophy; Progressive Supranuclear Palsy
Keywords: Parkinson disease; Multiple System Atrophy; MSA; Progressive Supranuclear Palsy; PSP; observational; biomarker
MeSH Terms: conditions — Parkinson Disease; Multiple System Atrophy; Supranuclear Palsy, Progressive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole Blood, serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The overall goal of PROBE is to evaluate the feasibility and potential utility of three markers (alpha-synuclein, transcriptomic profiles and olfactory function) to determine the risk or prognosis of PD.

DETAILED DESCRIPTION:
PROBE will test three biomarkers in PD subjects and controls to determine their feasibility and potential utility as markers of risk and prognosis for PD. This is a case control study, in which PD subjects will be compared to neurologically healthy controls and disease controls (MSA and PSP). The blood biomarker samples will be drawn once to evaluate blood alpha-synuclein levels as well as collection of lymphocyte mass for array analysis. Olfaction will be measured using the UPSIT for all subjects. The UPSIT will be conducted as part of PostCEPT for PD subjects and will only be repeated in this study for PD subjects in not done within 6 months. Control subjects may also choose to submit a blood specimen for processing and storage at the Coriell Institute for Medical Research, a research resource supported by the NINDS Human Genetics Resource Center.

Follow-up of the PD population over a 3-year period will allow us to evaluate the prognosis for important motor aspects of PD that will occur frequently in this cohort. These complications of PD include motor complications, postural instability, and non-motor impairment such as cognitive decline.

Healthy and disease control subjects may give permission at the Baseline visit to be contacted and followed in the previously established PSG FOUND study using mail and telephone contact to assess clinical status. Participation in the FOUND study provides another mechanism to maintain contact with subjects and collect supplemental data beyond that collected at the PROBE Baseline visit.

ELIGIBILITY:
Parkinson Disease Inclusion Criteria:

* Subject is participating in PostCEPT and meets UK brain bank criteria for PD
* Willing and able to provide informed consent

Healthy Control Inclusion Criteria:

* Spouse or non blood relative of the PD subject
* No known current diagnosis or history of a neurological disease
* MMSE score >27
* Age >45
* Willing and able to provide informed consent

Parkinsonism/Disease Control Inclusion Criteria (MSA and PSP)

* A diagnosis of Probable MSA based on Consensus Criteria OR Probable PSP based on NINDS-PSP Criteria
* Willing and able to provide informed consent

Exclusion Criteria for All Groups:

* Current use (within 7 days prior to Baseline Visit) of anticoagulants (e.g., warfarin or heparin)
* Known bleeding disorder (acquired or inherited)
* Known blood disorder (e.g. leukemia) or a history of anemia with a documented hematocrit <30
* Known pregnancy
* History of nasal trauma, sinusitis, or other nasal pathology that would interfere with smell testing

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic, spouses, PD patients from another trial
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2007-08; Primary Completion 2008-07 (Estimated)

PRIMARY OUTCOMES:
α-synuclein, transcriptomic profiles and olfactory function | Three years

SECONDARY OUTCOMES:
Unified Parkinson Disease Rating Scale (UPDRS) | Three Years
University of Pennsylvania Smell Identification Test (UPSIT) | Three Years

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Ravina, MD, Principal Investigator — University of Rochester
Locations (1):
- Parkinson Study Group, Rochester, New York, United States